CLINICAL TRIAL: NCT04611178
Title: DWI Cerebellar Infarct Volume as Predictor of Outcomes After Endovascular Treatment of Acute Basilar Artery Occlusion
Brief Title: Cerebellar Infarct Volume in Basilar Artery Stroke
Acronym: CIV-ABAO
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0596
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Ischemic Stroke
Keywords: MRI; Posterior fossa; Thrombectomy; Stroke
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CIV-ABAO: CIV-ABAO
  Interventions: Device: Mechanical thrombectomy

INTERVENTIONS:
Device: Mechanical thrombectomy — Stent retriever for treatment of cerebral arterial occlusions

SUMMARY:
Preprocedural predictors of outcome in patients with acute basilar artery occlusion (ABAO) who underwent endovascular treatment (EVT) remain controversial. Our aim was to analyze if pre-EVT diffusion-weighted images cerebellar infarct volume (CIV) was a predictor of 90-day outcomes.

DETAILED DESCRIPTION:
Acute basilar artery occlusion (ABAO) is a rare and devastating type of stroke. Endovascular treatment (EVT) is routinely performed in real-world practice, encouraged by guidelines from learned societies, and the recent result of the basilar artery international cooperation study (BASICS), a randomized controlled study.

ABAO may result in infarcts in the brainstem, cerebellar lobes, thalamus and subthalamic area, or occipitotemporal lobes. Previously, studies using the DWI Posterior-circulation Alberta Stroke Program Early CT (Pc-ASPECT) Score or brainstem score, for predicting outcome in patients with ABAO showed conflicting results. The rational for the brainstem scoring system was based on the anatomic architecture and the regional eloquence of brainstem, which may negatively influence functional outcome.

Nevertheless, one of the most significant and immediate dreaded complication, in patients with ABAO and cerebellar infarcts, is the development of a space-occupying edema. Due to the small volume of posterior fossa, cerebellar infarct with mass effect (CIMASS) contribute to a risk of catastrophic herniation with direct brainstem compression, hydrocephalus due to blockage of the fourth ventricle, or both. Up to 25% of patients with CIMASS deteriorate clinically resulting in morbidity and in mortality in 85% of patients without intervention. This potential risk of CIMASS, lead clinicians to strengthen clinical and radiological monitoring and modify therapeutic management with the recourse of live-saving suboccipital decompressive craniectomy (SDC), as recommended by learned societies.

Until now, little is known about predicting factors of outcomes in patients with ABAO treated by EVT and associated cerebellar infarct. In fact, there are no focusing research to assess if baseline cerebellar infarct volume (CIV) may correlate with 90-day clinical outcome and mortality, nor if such lesions would affect a reperfusion decision.

Using data of our prospective registry, the investigators analyzed consecutive MRI selected, endovascularly treated ABAO patients within the first 24h after symptom-onset. Using the initial Magnetic Resonance Imaging (MRI), baseline CIV was calculated in mL, on an apparent diffusion-coefficient map reconstruction (Olea sphere software).

CIV was analyzed in univariate and multivariable models as a predictor of 90-day functional independence (modified Rankin Scale [mRS] 0-2) and mortality. According to received operating characteristic (ROC) analysis, the optimal cut-off was determined by maximizing the youden index, to evaluate the prognostic value of CIV.

Our aim was to evaluate the frequency, the clinical, and radiological characteristics of cerebellar infarct, in a large cohort of ABAO selected by MRI prior to EVT, and to investigate the baseline CIV as a predictor of 90-day functional outcome and mortality.

ELIGIBILITY:
Inclusion criteria:

* patient with a clinical diagnosis of acute stroke in the posterior-circulation within 24 hours from symptom onset
* patient with a pertinent clinical deficit following physician evaluation (no NIHSS limit)
* acute basilar ischemia assessed on MRI matching clinical symptoms and including DWI; and
* ABAO confirmed by intra-arterial arteriography and treated using mechanical thrombectomy.

Exclusion criteria:

- Patients were excluded if they were ineligible for an MRI or ineligible for MT for the following reasons:

* prestroke modified Rankin Scale (mRS) score of >2
* life expectancy <3 months
* brainstem ischemia on DWI involving more than 80% of the area in axial view

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients >18 years, referred to our hospital, from January 2011 to October 2018, presenting acute basilar artery occlusion (ABAO) confirmed by magnetic resonance imaging treated by endovascular thrombectomy, with or without intravenous thrombolysis.
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2011-01-30 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Rate of Functional outcome at 90-day | 90 day
  90-day functional outcome A favorable outcome was defined as a 90-day mRS≤2.

SECONDARY OUTCOMES:
Mortality rate | 90 day
  Mortality and the cause of death at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Mourand, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC